CLINICAL TRIAL: NCT06036576
Title: Thyroid-Stimulating Hormone Levels and Recurrent Pregnancy Loss: Influence of Thyroxine Supplementation on Pregnancy Outcomes
Brief Title: Thyroxine Therapy for Recurrent Pregnancy Loss in Hypothyroid Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Kindy College of Medicine (Other)
Collaborators: Al-Elwyiah Maternity Teaching Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15 Al-KindyCM
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Early Pregnancy Loss; Thyroid Diseases
Keywords: Miscarriage; Hypothyroidism; Thyroid Stimulating Hormone; Thyroxin
MeSH Terms: conditions — Abortion, Habitual; Thyroid Diseases; Abortion, Spontaneous; Hypothyroidism | interventions — Thyroxine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thyroid Stimulating Hormone 2.5-4 mU/L (Active Comparator): This arm consists of participants who have experienced recurrent pregnancy loss in the first trimester and have TSH levels ranging between 2.5 mU/L and 4 mU/L. These participants will receive levothyroxine treatment of 1.6 micrograms per kg per day
  Interventions: Drug: Levothyroxine Pill
- Thyroid Stimulating Hormone more than 4 mU/L (Active Comparator): This arm consists of participants who have experienced recurrent pregnancy loss in the first trimester and have TSH levels more than 4 mU/L. These participants will receive levothyroxine treatment of 1.6 micrograms per kg per day
  Interventions: Drug: Levothyroxine Pill

INTERVENTIONS:
Drug: Levothyroxine Pill — all participants will receive levothyroxine treatment of 1.6 micrograms per kg per day early in the morning on empty stomach.
  Other Names: Euthyrox 50 Mcg Tablet, Merck

SUMMARY:
The goal of this clinical trial is to investigate the influence of thyroxine supplementation on pregnancy outcomes in women with varying levels of Thyroid-Stimulating Hormone (TSH), who have experienced recurrent pregnancy loss in the first trimester. The main questions it aims to answer are:

* Does thyroxine treatment improve pregnancy outcomes in women with TSH levels between 2.5 mU/L and 4 mU/L?
* Is the effect of thyroxine treatment different in women with TSH levels higher than 4 mU/L?

Participants will be grouped based on their TSH levels, into two groups - those with TSH levels between 2.5 mU/L and 4 mU/L, and those with TSH levels higher than 4 mU/L. They will then be given thyroxine treatment.

Researchers will compare these two groups to see if the pregnancy outcomes differ based on the different TSH levels and thyroxine treatment.

DETAILED DESCRIPTION:
This is a prospective clinical trial that aims to investigate the impact of thyroxine supplementation on the outcomes of pregnancies in women who have experienced recurrent pregnancy loss in the first trimester. The study will specifically focus on the role of Thyroid-Stimulating Hormone (TSH) levels in these outcomes.

Participants in the study will include women who have suffered recurrent pregnancy loss in the first trimester and exhibit varying levels of TSH. For the purpose of this research, these participants will be categorized into two groups based on their TSH levels: the first group will consist of women with TSH levels between 2.5 mU/L and 4 mU/L, and the second group will include those with TSH levels higher than 4 mU/L.

All participants will receive thyroxine treatment, with dosages and treatment plans as determined by their respective healthcare providers. The main purpose of this trial is to examine two key questions:

Does thyroxine treatment lead to improved pregnancy outcomes in women with TSH levels between 2.5 mU/L and 4 mU/L? How does the effect of thyroxine treatment on pregnancy outcomes differ in women with TSH levels higher than 4 mU/L? The primary outcomes of interest in this study will be pregnancy success rates, defined as a viable pregnancy beyond the first trimester. Secondary outcomes might include measurements such as gestational age at delivery, birth weight, and any complications that may arise during pregnancy.

This trial aims to provide valuable insights into the potential benefits of thyroxine treatment for women with varying levels of TSH who have experienced recurrent pregnancy loss. The results could contribute to the development of more effective treatment protocols and ultimately improve pregnancy outcomes for these women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 40 years old.
* Diagnosis of recurrent pregnancy loss, defined as two or more pregnancy losses in the first trimester.
* Confirmed thyroid function test results with TSH levels either between 2.5 and 4 or higher than 4.
* Willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Women who are currently taking thyroid medication before the study starts.
* Presence of other causes of recurrent pregnancy loss such as antiphospholipid syndrome, uterine abnormalities, genetic/chromosomal disorders, etc.
* Presence of other severe chronic diseases like heart disease, kidney disease, uncontrolled diabetes, etc.
* Known allergy or intolerance to thyroxine.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Pregnancy Success Rate | Assessed at the end of the first trimester (approximately 12 weeks of gestation) for each participant.
  The primary outcome measure will be the rate of successful pregnancies, defined as a viable pregnancy beyond the first trimester, among participants in each group. This outcome will be compared between the two groups to determine the impact of thyroxine treatment on successful pregnancies in women with varying levels of TSH.

SECONDARY OUTCOMES:
Gestational Age at Delivery | Assessed at the time of delivery for each participant.
  The gestational age at delivery will be recorded and compared between the two groups. This metric provides information about whether thyroxine treatment affects the timing of delivery in this population.
Birth Weight | Assessed at the time of delivery for each participant.
  The birth weight of the baby will be measured and compared between the two groups. This can provide further information on the potential effects of thyroxine treatment on pregnancy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Al-Musawi, C.A.B.O.G, Study Chair — Al-Kindy College of Medicine
Locations (1):
- AL-Elwiyah Maternity Teaching Hospital, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No